CLINICAL TRIAL: NCT06546995
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Effects of NMRA-323511 Among Healthy Elderly and Adults With Agitation Associated With Dementia Due to Alzheimer's Disease
Brief Title: Study to Evaluate the Effects of NMRA-323511 Among Healthy Elderly and Adults With Agitation Associated With Dementia Due to Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neumora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRA-323511-104
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease; Healthy Elderly
Keywords: Alzheimer's Disease; Agitation Associated Dementia; NMRA-323511
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: NMRA-323511 (Experimental)
  Interventions: Drug: NMRA-323511
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B: NMRA-323511 (Experimental)
  Interventions: Drug: NMRA-323511
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NMRA-323511 — Participants will receive NMRA-323511 orally.
  Arms: Part A: NMRA-323511; Part B: NMRA-323511
Drug: Placebo — Participants will receive matching placebo tablets orally.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
This study consists of 2 parts, Part A and Part B. Part A is a single center, randomized, double-blind, placebo-controlled cohort designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of NMRA-323511 among healthy elderly.

Part B is a multicenter, randomized, double-blinded, placebo-controlled, parallel-group cohort to evaluate the safety, tolerability, and efficacy of NMRA-323511 among adults with Agitation Associated with Dementia due to Alzheimer's Disease.

Part A consists of a Screening Period (up to 28 days), a 10-day Treatment Period, and a 10- day Follow-up clinic visit after last dose of study treatment.

Part B consists of a Screening Period (up to 28 days), an 8-week Treatment Period, and a 10-day Follow-up clinic visit after last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Healthy participants
* Age 65 to 80 years
* Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2 at the screening and check-in visit

Part B

* Participants aged 55 to 90 years
* Diagnosis of probable AD or Alzheimer's clinical syndrome according to the National Institute of Aging-Alzheimer's Association criteria at least 12 months prior to screening
* Agitation meets the International Psychogeriatric Association (IPA) consensus definition
* Mini-Mental State Examination (MMSE) score = 5 - 24 (mild to severe dementia) at screening

Exclusion Criteria:

Part A

* Participant is actively suicidal
* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit
* Diagnosis of epilepsy taking anticonvulsants for seizure control, history of seizures

Part B

* Dementia or memory impairment due to a reason other than AD
* Clinically significant neurologic disorder other than AD
* Have any clinically significant and uncontrolled medical condition

Note: Other protocol defined inclusion/exclusion criteria may apply

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability Assessments Based on Treatment Emergent Adverse Events (TEAEs) and Validated Clinical Scales | Up to 53 days
  An AE is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE). Clinically significant abnormalities in Clinical Laboratory Evaluations, ECGs, Vital Signs, Physical examinations, and Columbia Suicide Severity Rating Scale (C-SSRS) scores will be reported as TEAEs.
Part B: Safety and Tolerability Assessments Based on Treatment Emergent Adverse Events and Validated Clinical Scales | Up to Week 10
  An AE is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as a TEAE. Clinically significant abnormalities in Clinical Laboratory Evaluations, ECGs, Vital Signs, Physical examinations, and C-SSRS scores will be reported as TEAEs.
Part B: Change from Baseline to Week 8 on the Cohen-Mansfield Agitation Inventory (CMAI) Total Score | Baseline to Week 8
  The CMAI is a 29-item scale to assess the frequency of agitated behaviors. The 29 agitated behaviors are categorized into agitation factors, including aggressive behavior, physically non-aggressive behavior, and verbally agitated behavior. Each item is rated over the past 2 weeks on a 7-point scale ranging from "Never" (score of 1) to "Several times per hour" (score of 7). The CMAI total score is calculated as the sum of all 29 items and range from 29 (no agitation) to 203 (most severe agitation). A score >45 is commonly regarded as clinically significant agitation.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Neumora Investigator Site, Chandler, Arizona
  - Neumora Investigator Site, Tempe, Arizona
  - Neumora Investigator Site, Costa Mesa, California
  - Neumora Investigator Site, Lomita, California
  - Neumora Investigator Site, Walnut Creek, California
  - Neumora Investigator Site, Bradenton, Florida
  - Neumora Investigator Site, Greenacres City, Florida
  - Neumora Investigator Site, Hallandale, Florida
  - Neumora Investigator Site, Hialeah, Florida
  - Neumora Investigator Site, Miami, Florida
  - Neumora Investigator Site, Miami Springs, Florida
  - Neumora Investigator Site, Orlando, Florida
  - Neumora Investigator Site, Pembroke Pines, Florida
  - Neumora Investigator Site, Port Orange, Florida
  - Neumora Investigator Site, Atlanta, Georgia
  - Neumora Investigator Site, Honolulu, Hawaii
  - Neumora Investigator Site, Boise, Idaho
  - Neumora Investigator Site, Belmont, Massachusetts
  - Neumora Investigator Site, Troy, Michigan
  - Neumora Investigator Site, Toms River, New Jersey
  - Neumora Investigator Site, Brooklyn, New York
  - Neumora Investigator Site, East Syracuse, New York
  - Neumora Investigator Site, Charlotte, North Carolina
  - Neumora Investigator Site, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No